CLINICAL TRIAL: NCT00252785
Title: An 8-week, Randomised, Double Blind, Parallel-group, Multi-centre, Phase III Study Comparing the Efficacy and Safety of Symbicort® Turbuhaler® 160/4.5 µg Twice Daily and Pulmicort® Turbuhaler® 200 µg Twice Daily + Theolong® Tablet 200 mg Twice Daily in Japanese Patients With Asthma
Brief Title: Efficacy & Safety of Symbicort® TURBUHALER® 160/4.5 µg Twice Daily & Pulmicort® TURBUHALER® 200 µg Twice Daily + Theolong® Tablet 200 mg Twice Daily in Japanese Asthmatic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5890C00010
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Budesonide; Theophylline

INTERVENTIONS:
Drug: Budesonide/Formoterol
  Other Names: Symbicort
Drug: Budesonide
Drug: Theophylline

SUMMARY:
The primary objective of this study is to confirm the efficacy (superiority) of Symbicort® Turbuhaler® 160/4.5 µg twice daily for 8 weeks in comparison to Pulmicort® Turbuhaler® 200 µg twice daily + Theolong® tablet 200 mg twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma with a documented history of at least 6 months duration prior to Visit 1
* Prescribed daily use of an IGCS for >=12 weeks prior to Visit 1. The dose of IGCS must be 400 to 800 µg/day of Pulmicort® Turbuhaler® or corresponding dose of IGCS. The prescribed dose of IGCS should be constant for at least 4 weeks prior to Visit 1
* Prescribed daily use of sustained release theophylline for at least 8 weeks prior to Visit 1, or confirmed steady-state blood theophylline concentrations within the effective range (5-15 µg/mL) during 8 weeks prior to Visit 1. The prescribed dose of theophylline should be constant (400 mg/day) for at least 4 weeks prior to Visit 1

Exclusion Criteria:

* Any significant disease or disorder that may jeopardize the safety of the patient
* Respiratory infection, judged by the investigator(s) as an infection affecting the asthma, within 4 weeks prior to Visit 1
* Treatment with oral, parenteral or rectal GCS within 4 weeks prior to Visit 1

Additional inclusion and exclusion criteria will be evaluated by the Investigator

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 340
Dates: Start 2005-10; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Morning peak expiratory flow (mPEF)

SECONDARY OUTCOMES:
Patient reported outcomes regarding disease status (incl. evening PEF), collected via diaries
Forced expiratory volume in one second (FEV1)
Safety:
Adverse events (nature, incidence and severity)
Haematology, clinical chemistry and urinalysis
12-lead ECGs, blood pressure, pulse rate
- all variables assessed over the 8 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Symbicort Medical Science Director, MD, Study Director — AstraZeneca
Locations (43):
- Japan (43):
  - Research Site, Komaki, Aichi-ken
  - Research Site, Seto, Aichi-ken
  - Research Site, Asahi, Chiba
  - Research Site, Noda, Chiba
  - Research Site, Touon, Ehime
  - Research Site, Miyaodai, Fukuoka
  - Research Site, Gifu, Gifu
  - Research Site, Isesaki, Gunma
  - Research Site, Maebashi, Gunma
  - Research Site, Ōta, Gunma
  - Research Site, Ōwa, Gunma
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Chitose, Hokkaido
  - Research Site, Kitahiroshima, Hokkaido
  - Research Site, Obihiro, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Tomakomai, Hokkaido
  - Research Site, Morioka, Iwate
  - Research Site, Takamatsu, Kagawa-ken
  - Research Site, Kagoshima, Kagoshima-ken
  - Research Site, Kyoto, Kyoto
  - Research Site, Sendai, Miyagi
  - Research Site, Beppu, Ohita
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Okayama, Okayama-ken
  - Research Site, Tsukubo, Okayama-ken
  - Research Site, Kishiwada, Osaka
  - Research Site, Osaka, Osaka
  - Research Site, Oskasayama, Osaka
  - Research Site, Takatsuiki, Osaka
  - Research Site, Koshigaya, Saitama
  - Research Site, Minamisaitama, Saitama
  - Research Site, Arakawa City, Tokyo
  - Research Site, Chiyoda City, Tokyo
  - Research Site, Kodaira, Tokyo
  - Research Site, Nakano-ku, Tokyo
  - Research Site, Ōta-ku, Tokyo
  - Research Site, Shinagawa-ku, Tokyo
  - Research Site, Sumida City, Tokyo
  - Research Site, tabashi City, Tokyo
  - Research Site, Toyama, Toyama
  - Research Site, Ube, Yamaguchi
  - Research Site, Tochigi